CLINICAL TRIAL: NCT07194876
Title: A Survey Study Using the Ten-Group Robson Classification System to Evaluate Cesarean Section Rates and Maternal-Neonatal Outcomes in Assiut University Hospital and Assiut General Hospital
Brief Title: Robson Ten-Group Classification Study of Cesarean Section Rates in Assiut Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Elzahraa salah Sayed, Resident, Obstetric and Gynecology Department, Assiut University
Other Study IDs: AUN-OBGYN-RobsonCS-2026
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section; Maternal Health
Keywords: Robson Ten Group Classification; Cesarean Section Rate; Maternal Outcomes
MeSH Terms: interventions — saxagliptin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean Deliveries in Assiut Hospitals: Women who delivered by cesarean section at Assiut University Hospital or Assiut General Hospital dur
  Interventions: Other: No Intervention (subjects were previously treated with Onglyza®)

INTERVENTIONS:
Other: No Intervention (subjects were previously treated with Onglyza®) — no intervention

SUMMARY:
Cesarean section (C-section) rates have increased worldwide, and Egypt is among the countries with the highest rates. In some hospitals, more than half of all births are done by cesarean delivery. The World Health Organization (WHO) recommends using the "Robson Ten Group Classification System" to better understand and compare C-section rates.

This study will use the Robson classification system to evaluate the rate of cesarean deliveries in two hospitals in Assiut, Egypt: Assiut University Hospital and Assiut General Hospital. The study will collect information from medical records of women who delivered by cesarean section between January and December 2026.

The main goal is to identify which groups of women contribute most to the high C-section rate and to compare practices between the two hospitals. The study will also look at outcomes for both mothers and newborns. By doing this, we hope to provide useful information that can help improve obstetric care, reduce unnecessary cesarean deliveries, and improve health outcomes for mothers and babies in Egypt.

DETAILED DESCRIPTION:
Cesarean section (C-section) rates have risen dramatically worldwide, with Egypt showing one of the fastest increases, from 4.6% in 1992 to nearly 52% in 2014. Current national data indicate a rate of 51.8%, placing Egypt among the top three countries globally in C-section prevalence. This upward trend highlights an urgent need for systematic evaluation and targeted interventions.

In 2015, the World Health Organization (WHO) endorsed the Robson Ten Group Classification System (TGCS) as the international standard for assessing, monitoring, and comparing cesarean section rates. The TGCS categorizes all women into ten mutually exclusive and totally inclusive groups based on five basic obstetric characteristics: parity, previous cesarean section, onset of labor, gestational age, and fetal presentation. This approach allows for meaningful comparisons within and across institutions, identification of the main contributors to cesarean rates, and evaluation of adherence to evidence-based clinical practice.

Studies worldwide consistently report that Groups 5 (previous cesarean, single cephalic, ≥37 weeks), 2 (nulliparous, induced or elective), and 1 (nulliparous, spontaneous labor) are the major contributors to rising C-section rates. In Egypt, substantial variation exists across hospitals, with facility-specific C-section rates ranging from 22.9% to 94.3%. Previous studies at Assiut University Hospital showed an increase from 32% in 2008 to 38% in 2011, yet comparative analyses across different institutions remain scarce.

This prospective cross-sectional survey will be conducted between January and December 2026 in Assiut University Hospital and Assiut General Hospital. All women delivering by cesarean section during the study period will be eligible, with exclusion of incomplete medical records or deliveries before 28 weeks. The estimated sample size is 770 cases, accounting for incomplete records. Data will be extracted using a standardized Robson-based form and entered electronically.

Primary outcomes include:

Distribution of cesarean deliveries across Robson groups

Comparison of C-section rates within Robson groups between hospitals

Contribution of each Robson group to the overall C-section rate

Secondary outcomes include:

Maternal outcomes (mortality, complications, ICU admission, postpartum hemorrhage, length of stay)

Neonatal outcomes (birth weight, Apgar score, NICU admission, perinatal complications)

Analysis of C-section indications within Robson groups

Identification of potentially avoidable cesarean deliveries

Assessment of adherence to clinical guidelines

Data analysis will be performed using SPSS v29.0. Statistical methods include descriptive analysis, chi-square tests, Fisher's exact tests, t-tests, logistic regression, and propensity score matching. A p-value <0.05 will be considered significant.

The results of this study will provide evidence on institutional differences in cesarean section practices in Assiut, inform local health policies, and support interventions aimed at optimizing the use of cesarean delivery to improve maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who delivered by cesarean section at Assiut University Hospital or Assiut General Hospital during the study period (January-December 2026).

Gestational age ≥ 28 weeks.

Complete medical records available.

Exclusion Criteria:

* Vaginal deliveries.

Cesarean deliveries before 28 weeks of gestation.

Incomplete or missing medical records.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women delivering by cesarean section at Assiut University Hospital and Assiut General Hospital in Assiut, Egypt, between January and December 2026. Data will be collected from medical records and classified using the Robson Ten Group Classification System.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of cesarean deliveries by Robson Ten Group Classification | January 2026 - December 2026
  Proportion of cesarean section deliveries categorized into the ten Robson groups, calculated as a percentage of total cesarean deliveries. The main objective is to identify the groups contributing most to the overall cesarean section rate.

SECONDARY OUTCOMES:
Comparison of cesarean section rates within Robson groups between hospitals | January 2026 - December 2026
  Rate and relative contribution of each Robson group will be compared between Assiut University Hospital and Assiut General Hospital.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 3. World Health Organization. Robson classification: implementation manual. Geneva: WHO; 2017.
- [Background] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Background] Elnakib S, Abdel-Tawab N, Orbay D, Hassanein N. Medical and non-medical reasons for cesarean section delivery in Egypt: a hospital-based retrospective study. BMC Pregnancy Childbirth. 2019 Nov 8;19(1):411. doi: 10.1186/s12884-019-2558-2. PMID 31703638